CLINICAL TRIAL: NCT06912009
Title: Evaluation of the Duration of Obtaining Curative Anticoagulation in Patients With Clinically Significant Pulmonary Embolism in an Intensive Care Unit
Brief Title: Duration of Therapeutic Anticoagulation in Patients With Pulmonary Embolism
Acronym: ACEP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9373
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Curative Anticoagulation; Fibrinolytic therapy; Thrombectomy
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current management of intermediate- and high-risk pulmonary embolism is primarily based on curative subcutaneous or intravenous anticoagulation, with or without systemic fibrinolytic therapy or thrombectomy. Initial treatment with low-molecular-weight heparin (LMWH) or fondaparinux is preferred over unfractionated heparin (UFH) due to their lower risk of serious bleeding and heparin-induced thrombocytopenia (HIT). UFH treatment is reserved for patients at risk of hemodynamic instability, renal failure with a GFR < 30 ml/min, or obesity. Biological monitoring of anticoagulation efficacy can be performed by measuring the activated partial thromboplastin time (aPTT), as recommended by the European Society of Cardiology (ESC), or by measuring the antiXa activity of heparin, which has been shown to be beneficial in numerous studies. It is generally accepted that this anticoagulation should be initiated at a curative dose as early as possible, as this reduces in-hospital mortality and 30-day mortality. However, few studies have examined the impact of the time to achieve effective anticoagulation, and those that have done so have only done so in patients with high-risk pulmonary embolism or have based their anticoagulation monitoring on aPTT and not on antiXa activity.

The proposed study aims to evaluate the time to obtain effective anticoagulation and its impact on mortality, thromboembolic recurrence and the occurrence of serious bleeding in patients with clinically significant pulmonary embolism, hospitalized in an intensive care unit as well as the factors that may influence this time. It will also allow to compare the practices of the studied center in terms of initial anticoagulation dose delivered, the initiation or not of a bolus and methods of monitoring anticoagulation with the literature in order to allow an improvement in patient care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Hospitalized in the intensive care unit of Hautepierre Hospital (Strasbourg University Hospitals UF 6250) between January 1, 2014, and December 31, 2023
* With a diagnosis of pulmonary embolism confirmed by a thoracic CT angiogram, a thoracoabdominopelvic CT scan, or a lung scan
* Having received anticoagulation with curative-dose unfractionated heparin

Exclusion Criteria:

* Subjects who have expressed objection to the reuse of their data for scientific research purposes. - Patients diagnosed with pulmonary embolism prior to admission to the intensive care unit and for whom we cannot precisely determine the start date of anticoagulation (precision estimated to the nearest hour).
* Pulmonary embolism not confirmed by contrast imaging (CT angiography)
* Patients who have not received curative anticoagulation (contraindication)
* Patients already receiving curative anticoagulation with UFH at the time of diagnosis
* Patients with low-risk pulmonary embolism defined by an sPESI score of 0
* Subject under court protection, guardianship, or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) hospitalized in the intensive care unit of Hautepierre Hospital (Strasbourg University Hospitals UF 6250) between January 1, 2014, and December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the time to effective anticoagulation with HNF in the treatment of high-risk and intermediate-risk pulmonary embolism in an intensive care unit. | Up to 10 years
  Mean time to achieve effective anticoagulation, defined as the mean time between the initiation of curative anticoagulation and the first antiXa activity value greater than 0.3 units/ml in the case of antiXa monitoring, or an aPTT ratio > 2 in the case of aPTT monitoring. In the case of monitoring by both aPTT ratio and antiXa activity, the antiXa activity value will be preferred.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Médicale - CHU de Strasbourg - France, Strasbourg, France